CLINICAL TRIAL: NCT03970200
Title: A Phase II, Randomized Trial to Evaluate the Safety and Efficacy of Fecal Microbiota Transplantation Using the Penn Microbiome Therapy Products for Severe or Severe-Complicated/Fulminant Clostridium Difficile Infection
Brief Title: Penn Microbiome Therapy (PMT) for Severe-Clostridium Difficile Infection (CDI)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Administrative reasons.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 832962
Record Dates: First submitted 2019-04-17; First posted 2019-05-31 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Severe Clostridium Difficile Infection; Severe-Complicated/Fulminant Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Randomized, open label, comparative
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- No investigational product (Active Comparator): Participants who receive the antibiotics usually prescribed for C diff infection.
  Interventions: Drug: Antibiotics
- Upper gastrointestinal Fecal Microbiota Transplantation (Experimental): Participants who receive the antibiotics usually prescribed for C diff infection, along with PMT that is given by mouth in capsules or through a tube that goes into your stomach/intestines if you already have one (upper delivery). You will not be assigned to this group if you cannot take any medications either by mouth or through a tube safely, as determined by your doctor
  Interventions: Drug: Penn Microbiome Therapy - 002; Drug: Penn Microbiome Therapy - 003; Drug: Antibiotics
- Lower gastrointestinal Fecal Microbiota Transplantation (Experimental): Participants who receive the antibiotics usually prescribed for C diff infection, along with PMT that is given through the rectum by an enema (lower delivery).
  Interventions: Drug: Penn Microbiome Therapy - 001; Drug: Antibiotics

INTERVENTIONS:
Drug: Penn Microbiome Therapy - 001 — Fecal Microbiota for Transplant, enema product
  Other Names: PMT-001
  Arms: Lower gastrointestinal Fecal Microbiota Transplantation
Drug: Penn Microbiome Therapy - 002 — Fecal Microbiota for Transplant, suspension product
  Other Names: PMT-002
  Arms: Upper gastrointestinal Fecal Microbiota Transplantation
Drug: Penn Microbiome Therapy - 003 — Fecal Microbiota for Transplant, capsule product
  Other Names: PMT-003
  Arms: Upper gastrointestinal Fecal Microbiota Transplantation
Drug: Antibiotics — Standard of care antibiotics

SUMMARY:
This is a randomized, open label, comparative, Phase II study to determine whether fecal microbiota transplant using Penn Microbiome Therapy products helps standard therapy to treat severe Clostridium difficile infection (C diff).

ELIGIBILITY:
Inclusion Criteria:

* 1. One or more episodes of CDI with symptoms including bowel movements altered in frequency or consistency from baseline.
* 2. Stool test positive for Clostridium difficile by enzyme immunoassay (EIA) by FDA-cleared assay within 7 days prior to enrollment.
* 3. Age ≥ 18 years
* 4. Meets any one of the listed criteria for severe or severe-complicated/fulminant disease within 72 hours of enrollment.
* 5. Receiving antibiotic treatment for S/SC(Severe-complicatedcategory)/F-CDI per current Infectious Diseases Society of America(IDSA) guidelines.

Enrollment criteria details:

* 1. Must either meet ≥1 criteria in severe category or in severe complicated category to be enrolled
* 2. If the subject meets criteria in both categories, stratify to the higher severity category (severe complicated)
* 3. Detailed enrollment criteria definitions:
* a. white blood cells (WBC) ≥15,000 cells/uL - if any value in the time period meets this definition
* b. Hypotension with systolic blood pressure sustained < 90mmHg for three or more hours or requiring vasopressors (epinephrine, norepinephrine, phenylephrine, or vasopressin)
* c. Acute kidney injury - increase in serum creatinine level by ≥50% or new dialysis initiation
* i. If a baseline serum creatinine value is not available, acute kidney injury will be defined as a serum creatinine >1.5 mg/dL
* d. Temperature ≥38.5 °C or <35.6°C - one value needed in time period -
* e. Ileus, bowel dilation or megacolon
* i. Ileus: If noted in any provider documentation or problem list (search words "ileus") OR
* ii. If the words "dilated" "dilation" or "ileus" are noted in a radiology report on intestines/colon, or if "megacolon" noted
* f. Lactate >2.2 mmol/L - if any value in the time period meets this definition
* g. Systemic inflammatory response syndrome(SIRS) criteria
* i. Heart rate > 90 beats per minute
* ii. Respiratory rate > 20 breaths per minute or PaCO2 < 32 mmHg
* iii. Temperature >38ºC or <36ºC
* iv. WBC > 12,000 cells/uL, <4,000 cells/uL, or >10% immature (band) forms

Exclusion Criteria:

* 1. Evidence of colon/small bowel perforation at the time of study screening.
* 2. Goals of care are directed to comfort rather than curative measures.
* 3. Moderate (ANC < 1000 cells/uL) or severe (ANC < 500 cells/uL) neutropenia.
* 4. Known food allergy that could lead to anaphylaxis.
* 5. Pregnancy
* a. For subjects of childbearing potential (ages 18 to 55), the subject must have a negative urine pregnancy test within 48 hours of consent and no more than 48 hours prior to first product administration.
* 6 Receipt of Fecal Microbiota Transplantation (FMT) or enrollment in a clinical trial for FMT within the last 3 months.
* 7 COVID-19 infection, as defined by a positive nucleic acid or antigen test within the prior 14 days and symptoms consistent with COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-11-21 (Actual); Study Completion 2022-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ebbing Lautenbach, MD, MPH, MSCE, Principal Investigator — Division of Infectious Diseases, Department of Medicine, University of Pennsylvania
Locations (1):
- Hospital of the Univeristy of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Upper Gastrointestinal Fecal Microbiota Transplantation: Participants who receive the antibiotics usually prescribed for C diff infection, along with Penn Microbiome Therapy (PMT) that is given by mouth in capsules or through a tube that goes into your stomach/intestines if you already have one (upper delivery). You will not be assigned to this group if you cannot take any medications either by mouth or through a tube safely, as determined by your doctor
  Penn Microbiome Therapy - 002: Fecal Microbiota for Transplant, suspension product
  Penn Microbiome Therapy - 003: Fecal Microbiota for Transplant, capsule product
  Antibiotics: Standard of care antibiotics
Period: Overall Study
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation
Started | 5 | 4 | 6
Completed | 3 | 2 | 4
Not Completed | 2 | 2 | 2
Not completed — Death | 2 | 2 | 1
Not completed — Subject re-enrolled into Upper GI | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation | Total
Number analyzed (Participants) | 5 | 4 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 3 | 3
  >=65 years | 5 | 4 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 7
  Male | 3 | 3 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3
  White | 2 | 3 | 5 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Resolution of Symptoms After Treatment With One of the PMT Suite of Products.
Description: The outcome will be satisfied when the subject is discharged from the hospital (not to hospice or palliative care) or, while the subject remains hospitalized, when the following criteria are met for 72 hours:
  * If radiology study or studies performed, ileus/dilation/megacolon either not noted or noted as resolved
  * Ileus/megacolon either noted as resolved by any provider documentation or not noted
  * White Blood Cells (WBC) <15,000 cells/uL
  * Serum creatinine decreased, unchanged, or increased by ≤0.2 mg/dL over 72 hours (if not receiving continuous renal replacement therapy (CRRT) or hemodialysis (HD))
  * Lactate ≤2.2 mmol/L (if measured by clinical care team)
  * No vasopressors used (including epinephrine, norepinephrine, phenylephrine, or vasopressin)
  * Temperature <38.5 °C and ≥35.6°C
  * < 8 bowel movements per day and < 600 mL unformed stool (if volume recorded)
  * Meeting fewer than 3 systemic inflammatory response syndrome (SIRS) criteria
Time Frame: 3 Days
Measure: Count of Participants; unit: Participants
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation
Number analyzed (Participants) | 5 | 4 | 6
Participants | 4 | 3 | 5

2. Secondary Outcome: All-cause Mortality at 30 Days Following Last Fecal Microbiota Transplantation (FMT)
Description: Number of deaths within 30 days of the last FMT
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation
Number analyzed (Participants) | 5 | 4 | 6
Participants | 1 | 2 | 1

3. Secondary Outcome: All-cause Mortality at 60-days Following Last FMT
Description: Number of deaths within 60 days of the last FMT
Time Frame: 60 Days
Measure: Count of Participants; unit: Participants
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation
Number analyzed (Participants) | 5 | 4 | 6
Participants | 1 | 2 | 1

4. Secondary Outcome: Colectomy or Diverting Ileostomy Within 30 Days After Last FMT
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation
Number analyzed (Participants) | 5 | 4 | 6
Participants | 0 | 0 | 0

5. Secondary Outcome: Cumulative Days of Hospitalization From Enrollment Until 30 Days After FMT
Time Frame: 30 Days
Measure: Median (Full Range); unit: days
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation
Number analyzed (Participants) | 5 | 4 | 6
days | 13 [6 to 16] | 8 [4 to 13.5] | 14 [4 to 16]

6. Secondary Outcome: Cumulative Days in Intensive Care Unit From Enrollment Until 30 Days After Last FMT
Time Frame: 30 Days
Measure: Median (Full Range); unit: days
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation
Number analyzed (Participants) | 5 | 4 | 6
days | 0 [0 to 0] | 0 [0 to 4.5] | 0 [0 to 2]

7. Secondary Outcome: Bacteremia From Enrollment Until 30 Days After Last FMT
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation
Number analyzed (Participants) | 5 | 4 | 6
Participants | 0 | 0 | 0

8. Secondary Outcome: Repeat Hospital Admission Within 60 Days of Discharge From Index Hospitalization
Time Frame: 60 Days
Measure: Count of Participants; unit: Participants
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation
Number analyzed (Participants) | 5 | 2 | 6
Participants | 2 | 1 | 3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | No Investigational Product | Upper Gastrointestinal Fecal Microbiota Transplantation | Lower Gastrointestinal Fecal Microbiota Transplantation
All-Cause Mortality (participants affected / at risk) | 2/5 | 2/4 | 1/6
Serious Adverse Events (participants affected / at risk) | 3/5 | 3/4 | 4/6
Other Adverse Events (participants affected / at risk) | 4/5 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Investigational Product (N=5) | Upper Gastrointestinal Fecal Microbiota Transplantation (N=4) | Lower Gastrointestinal Fecal Microbiota Transplantation (N=6)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Death NOS (General disorders) | 2 (2) | 2 (2) | 1 (1)
Edema limbs (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Adenocarcinoma
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Left lung adenocarcinom
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Investigational Product (N=5) | Upper Gastrointestinal Fecal Microbiota Transplantation (N=4) | Lower Gastrointestinal Fecal Microbiota Transplantation (N=6)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Splenomegaly
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — Thrombocytopenia and Leukopenia
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Endocrine disorders - Other (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) — Diabetes
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (5) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations-Other (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) — Bacteriuria
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) — Glioblastoma (progression)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Genital edema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders-Other (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — Squamous cell carcinoma
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03970200/Prot_SAP_000.pdf